CLINICAL TRIAL: NCT02566278
Title: Determination of Upper Airway Collapsibility During Routine CPAP Titration
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Data collection has been halted. We are not recruiting any more subjects.
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Robert L. Owens, Assistant Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UCSD151355
Record Dates: First submitted 2015-09-26; First posted 2015-10-02 (Estimated); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive Sleep Apnea; Pcrit; Upper airway collapsibility
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Obstructive Sleep Apnea (Experimental): Upper airway collapsibility (passive Pcrit) will be measured using both clinically available equipment and research equipment in patients with obstructive sleep apnea (OSA) and stable on treatment of continuous positive airway pressure (CPAP) > 3 months to verify the Pcrit measurement obtained by the clinical equipment.
  Interventions: Other: Upper airway collapsibility (Pcrit)

INTERVENTIONS:
Other: Upper airway collapsibility (Pcrit) — To measure passive Pcrit, patients sleep with a mask over their nose or nose and mouth, and CPAP is applied using a custom made machine that can rapidly change mask pressures in research setting. The idea is that rapid changes in airway pressure produce a clear step change in airflow that will be observed quickly. In contrast, during clinical titrations, the CPAP machines change pressure much more slowly to help promote patient comfort. Passive Pcrit will be measured using both research and clinical equipment in the same patients and the Pcrit result using clinical CPAP titration equipment will be compared to the gold standard: Pcrit measurement done through research equipment that changes CPAP pressure rapidly.

SUMMARY:
The investigators hypothesis is that upper airway collapsibility (Pcrit) in patients with obstructive sleep apnea (OSA) can be measured using equipment found in the clinical sleep laboratory and these Pcrit measurements obtained using clinical sleep laboratory equipment is comparable to those obtained using research equipment. OSA is a common disease characterized by repetitive collapse of the upper airway during sleep, leading to hypoxemia and arousals, and which has important neurocognitive and cardiovascular consequences. The single most important factor in the development of OSA is upper airway collapsibility: those with a more collapsible upper airway tend to have OSA while those with a stiffer upper airway do not. The gold standard treatment for OSA is continuous positive airway pressure (CPAP), which acts by stenting open the collapsible airway. Upper airway collapsibility can be measured during sleep by changing the CPAP level and assessing the change in inspiratory flow through the upper airway. Although technically feasible, these measurements are typically only undertaken in research laboratories with specialized equipment. The purpose of this study is to measure upper airway collapsibility using clinically available (i.e. equipment found in a clinical sleep laboratory) equipment only. If successful, upper airway collapsibility could be routinely measured in clinical practice, which could help inform treatment decisions and help individualize therapy for OSA.

DETAILED DESCRIPTION:
OSA is defined by total or partial intermittent collapse of the upper airway, resulting in nocturnal hypoxemia and arousals from sleep. OSA is incredible common and has important cardiovascular (e.g. hypertension, coronary artery disease, stroke, atrial fibrillation) and neurocognitive consequences (e.g. depression, motor vehicle accidents). Thus, OSA results in significant morbidity and mortality and a substantial economic burden. The best studied treatment of OSA is continuous positive airway pressure (CPAP), which effectively stents the upper airway open, however, many patients are not able to tolerate it. Other treatments are available, such as oral appliances or upper airway surgery, however these are much more variable in their effectiveness.

Although other factors are important, the most important factor in OSA pathogenesis is upper airway collapsibility. The upper airway collapsibility can be determined during sleep when patients with OSA are on CPAP. The CPAP level is decreased until flow limitation and finally collapse is achieved. The pressure at which the airway collapses is called the pharyngeal critical closing pressure, or Pcrit. When measured in research laboratories, the Pcrit correlates with OSA severity. Subjects with a high Pcrit (e.g. 5cm of water pressure) typically have severe OSA, while those with a lower Pcrit (e.g. 2cm of water pressure) have mild OSA, and those with a negative Pcrit (e.g. -4cm of water, the airway must be sucked closed to collapse) typically have no disease. The Pcrit may also have important implications for treatment. For example, patients with OSA and a very high Pcrit may require CPAP, however, those with a lower or slightly negative Pcrit might be successfully treated by an oral appliance. Thus, knowledge of the Pcrit might be useful in clinical practice, but it is rarely measured outside of the research lab.

To measure Pcrit, patients sleep with a mask over their nose or nose and mouth, and CPAP is applied using a custom made machine that can rapidly change mask pressures. The idea is that rapid changes in airway pressure produce a clear step change in airflow that will be observed quickly. In contrast, during clinical titrations, the CPAP machines change pressure much more slowly to help promote patient comfort. The goal of this research is to determine whether these slower pressure changes could still be used to gather useful information about upper airway collapsibility.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of OSA and stable on CPAP treatment > 3 months

Exclusion Criteria:

* Pregnancy
* Currently smoking
* Any respiratory disorder other than OSA or well controlled asthma
* Medications known to affect respiratory function (e.g. opioids, benzodiazepines, etc)

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-10-20 (Actual); Primary Completion 2016-07-25 (Actual); Study Completion 2016-07-25 (Actual)

PRIMARY OUTCOMES:
Passive critical closing pressure (Pcrit) | Baseline
  Upper airway collapsibility, as measured by critical closing pressure (Pcrit), defined as the maximum nasal pressure at which the upper airway occludes.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Owens, MD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, San Diego, California, United States

REFERENCES:
- [Background] Malhotra A, Orr JE, Owens RL. On the cutting edge of obstructive sleep apnoea: where next? Lancet Respir Med. 2015 May;3(5):397-403. doi: 10.1016/S2213-2600(15)00051-X. Epub 2015 Apr 14. PMID 25887980
- [Background] Wei T, Erlacher MA, Grossman P, Leitner EB, McGinley BM, Patil SP, Smith PL, Schneider H, Schwartz AR, Kirkness JP. Approach for streamlining measurement of complex physiological phenotypes of upper airway collapsibility. Comput Biol Med. 2013 Jun;43(5):600-6. doi: 10.1016/j.compbiomed.2012.12.006. Epub 2013 Mar 18. PMID 23517555
- [Background] Owens RL, Edwards BA, Eckert DJ, Jordan AS, Sands SA, Malhotra A, White DP, Loring SH, Butler JP, Wellman A. An Integrative Model of Physiological Traits Can be Used to Predict Obstructive Sleep Apnea and Response to Non Positive Airway Pressure Therapy. Sleep. 2015 Jun 1;38(6):961-70. doi: 10.5665/sleep.4750. PMID 25515107
- [Background] Eckert DJ, White DP, Jordan AS, Malhotra A, Wellman A. Defining phenotypic causes of obstructive sleep apnea. Identification of novel therapeutic targets. Am J Respir Crit Care Med. 2013 Oct 15;188(8):996-1004. doi: 10.1164/rccm.201303-0448OC. PMID 23721582
- [Background] Owens RL, Malhotra A, Eckert DJ, White DP, Jordan AS. The influence of end-expiratory lung volume on measurements of pharyngeal collapsibility. J Appl Physiol (1985). 2010 Feb;108(2):445-51. doi: 10.1152/japplphysiol.00755.2009. Epub 2009 Nov 25. PMID 19940097